CLINICAL TRIAL: NCT04402476
Title: Skin Sensitisation Test (Modified Draize-95) to Support a Low Dermatitis Potential Claim
Brief Title: Skin Sensitisation (Modified Draize-95 Test)
Acronym: MDT-95
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT. Medisafe Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR-MDT-02-19-19-PT.MT
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Skin Sensitisation

STUDY DESIGN:
Intervention Model Description: Powder Free Polychloroprene Surgical Glove, Sterile. Low Dermatitis Potential, tested for use with chemotherapy drugs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device and Control (Experimental): Device:
  Powder Free Polychloroprene Surgical Gloves, Sterile. Low Dermatitis Potential, Tested for use with Chemotherapy Drugs.
  Approximately 2cm x 2cm square positioned to ensure that the inside portion of the test material maintained skin contact.
  Positive Control:
  0.4% Sodium Lauryl Sulfate (SLS) Dose. 0.2 ml
  Interventions: Device: Powder Free Polychloroprene Surgical Gloves, Sterile. Low Dermatitis Potential, tested for use with Chemotherapy drugs.

INTERVENTIONS:
Device: Powder Free Polychloroprene Surgical Gloves, Sterile. Low Dermatitis Potential, tested for use with Chemotherapy drugs. — Approximately 2cm x 2cm square positioned to ensure that the inside portion of the test material maintained skin contact.

SUMMARY:
Skin Sensitization Test (Modified Draize-95) to Support a Low Dermatitis Potential Claim for a Powder Free Polychloroprene Surgical Gloves, Sterile. To evaluate whether residual chemical additives at a level on the gloves that may induce type IV allergy to the unsensitized general user population when using polychloroprene based surgical gloves

DETAILED DESCRIPTION:
1. To evaluate whether residual chemical additives at a level that may induce Type IV allergy in the unsensitized general user population are present in a finished Polychloroprene Rubber Containing Medical Device, Powder Free Polychloroprene Surgical Gloves, Sterile. (CR-SG-140-AF-WH)
2. To meet requirements for claim: This product demonstrated reduced potential for sensitizing users to chemical additives as described in Guidance for Industry and FDA Staff- Medical Glove Guidance Manual. Supporting Test Data: A negative skin sensitization test (Modified Draize-95 Test) on a minimum of 200 non-sensitized human subjects.

ELIGIBILITY:
Inclusion Criteria:

* The test subjects are normal volunteers who have documented informed consent and have not participated in other voluntary testing for at least 30 days.
* Age of the test subjects ranged from 18 to 65 years.
* Efforts are made to provide racial and gender diversity of the test subjects that reasonably reflects the general user population in the US

Exclusion Criteria:

* The test subjects with any visible skin disease that might be confused with skin reactions caused by the test material.
* The test subjects with any indication of existing Type I allergy to natural rubber proteins.
* The test subjects who have used corticosteroids, either systemically or topically on the potential test site, two weeks before testing.
* Test subjects who have received endogenous or exogenous immunosuppressive treatments (or prolonged sun exposure).
* All subjects who are pregnant or become pregnant during the study.
* All lactating women,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 104 female (50%) and 104 male (50%)
Enrollment: 208 (Actual)
Dates: Start 2019-11-23 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Induction Phase | 24 days
  Irritation scored by Erythemal Scoring Scale,
  Basic Score - Description:
  0 - No visible reaction.
  0.5 - Doubtful or Negligible Erythema Reaction.
  1.0 - Mild or just perceptible macular erythema reaction in a speckled / follicular, patchy or confluent pattern (slight pinking).
  2.0 - Moderate erythema reaction in a confluent pattern (definite redness).
  3.0 - Strong or brisk erythema reaction that may spread beyond the test site.
Challenge Phase | 48 hours
  Irritation scored by Erythemal Scoring Scale,
  Basic Score - Description :
  0 - No visible reaction.
  0.5 - Doubtful or Negligible Erythema Reaction.
  1.0 - Mild or just perceptible macular erythema reaction in a speckled / follicular, patchy or confluent pattern (slight pinking).
  2.0 - Moderate erythema reaction in a confluent pattern (definite redness).
  3.0 - Strong or brisk erythema reaction that may spread beyond the test site.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Saadiah Sulaiman, Dermatologist, MBBCh, MMED, Study Director — Makmal Bioserasi & Klinikal, Healthmedic Research Sdn. Bhd.
Locations (1):
- Makmal Bioserasi & Klinikal, Healthmedic Research Sdn. Bhd., Kuala Lumpur, Cheras, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Foy V, Weinkauf R, Whittle E, Basketter DA. Ethnic variation in the skin irritation response. Contact Dermatitis. 2001 Dec;45(6):346-9. doi: 10.1034/j.1600-0536.2001.450605.x. PMID 11846750
- [Result] Kompaore F, Tsuruta H. In vivo differences between Asian, black and white in the stratum corneum barrier function. Int Arch Occup Environ Health. 1993;65(1 Suppl):S223-5. doi: 10.1007/BF00381346. PMID 8406931
- [Result] Robinson MK. Population differences in acute skin irritation responses. Race, sex, age, sensitive skin and repeat subject comparisons. Contact Dermatitis. 2002 Feb;46(2):86-93. doi: 10.1034/j.1600-0536.2002.460205.x. PMID 11918601
- See also: Medical Glove Guidance Manual — http://www.fda.gov/downloads/medicaldevices/deviceregulationandguidance/guidancedocuments/ucm428191.pdf
- See also: Guidance for Industry and FDA Reviewers/Staff: Premarket Notification [510(k)] Submissions for Testing for Skin Sensitization To Chemicals In Natural Rubber Products. — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/premarket-notification-510k-submissions-testing-skin-sensitization-chemicals-natural-rubber-products